CLINICAL TRIAL: NCT00445120
Title: Multicenter, Randomised, Double Masked, Controlled Studies on the Efficacy of Lactobacillus Rhamnosus GG Treatment in Preventing Vernal Keratoconjunctivitis VKC) Relapses.
Brief Title: Lactobacillus Rhamnosus GG Oral Treatment Efficacy on Vernal Keratoconjunctivitis Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Collaborators: University of Genova (Other); University of Padova (Other)
Responsible Party: Stefano Bonini, University of Rome Campus Bio-Medico
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LACTO2; Eudract number 2007-000209-31
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: Vernal keratoconjunctivitis; probiotic; Lactobacillus Rhamnosus GG; Children; Clinical trial
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Lactobacillus Rhamnosus GG
- 2 (Placebo Comparator)
  Interventions: Drug: placebo (sugar)

INTERVENTIONS:
Drug: Lactobacillus Rhamnosus GG — patients are treated with oral Lactobacillus Rhamnosus GG once daily for six months
  Arms: 1
Drug: placebo (sugar) — Placebo will be administered to patients once daily for six months
  Arms: 2

SUMMARY:
This interventional study aims to evaluate the efficacy of oral administration of Lactobacillus Rhamnosus GG in preventing relapses of ocular inflammation in Vernal Keratoconjunctivitis (VKC) patients.

DETAILED DESCRIPTION:
Vernal keratoconjunctivitis (VKC) is a chronic allergic disease, characterised by ocular surface inflammation lasting all year with seasonal relapses. Active phases of VKC are characterised by intense ocular symptoms and require treatment with topical steroids to control inflammation and corneal damage. To date, safe and effective therapies in preventing relapses of VKC are not available. Recently, the use of oral administration of probiotics for allergic diseases have been proposed. No data are available on the effects of probiotics on ocular allergies. This multicenter, double-masked, randomised, controlled clinical trial will allow to obtain more data on the efficacy of oral treatment with Lactobacillus Rhamnosus GG in patients affected by VKC. Patients with VKC will be treated with Lactobacillus Rhamnosus GG or placebo in addition to ketotifen fumarate 0.025% eye drops (standard treatment). The number of relapses per year, signs and symptoms of the disease, total symptom score (TSyS), total sign score (TSS), biochemical and molecular parameters will be evaluated at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of VKC performed on the basis of personal and family history of systemic allergic diseases, clinical examination (presence of conjunctival tarsal and/or limbal papillae) and presence of eosinophils in the conjunctival scraping.

Exclusion Criteria:

* Contact lens wearers,
* Patients affected by other ocular diseases,
* Patients subjected to ocular surgery in the preceding 6 months,
* Patients under eye drop or systemic treatments for other diseases,
* Patients enrolled in experimental trials in the preceding 6 months.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate a difference in the number of relapses of ocular inflammation for year between Lactobacillus Rhamnosus GG and placebo treated groups. Relapses will be defined as at least 100% increase of the sum of hyperemia, | 2 years

SECONDARY OUTCOMES:
Differences of specific symptoms and signs, TSyS, TSS, Quick questionnaire subscales,biochemical and molecular parameters will be evaluated at baseline, after 1, 3 and 6 months of treatment and after 1 month of treatment discontinuation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bonini, MD, Study Director — University Campus Bio-Medico
Locations (3):
- Italy (3):
  - University of Genova, Genova
  - University of Padua, Padua
  - University Campus Bio-Medico, Rome

REFERENCES:
- [Background] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Background] Kalliomaki M, Salminen S, Poussa T, Arvilommi H, Isolauri E. Probiotics and prevention of atopic disease: 4-year follow-up of a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1869-71. doi: 10.1016/S0140-6736(03)13490-3. PMID 12788576
- [Background] Boyle RJ, Tang ML. The role of probiotics in the management of allergic disease. Clin Exp Allergy. 2006 May;36(5):568-76. doi: 10.1111/j.1365-2222.2006.02472.x. PMID 16650040
- [Background] Peng GC, Hsu CH. The efficacy and safety of heat-killed Lactobacillus paracasei for treatment of perennial allergic rhinitis induced by house-dust mite. Pediatr Allergy Immunol. 2005 Aug;16(5):433-8. doi: 10.1111/j.1399-3038.2005.00284.x. PMID 16101937
- [Background] Viljanen M, Savilahti E, Haahtela T, Juntunen-Backman K, Korpela R, Poussa T, Tuure T, Kuitunen M. Probiotics in the treatment of atopic eczema/dermatitis syndrome in infants: a double-blind placebo-controlled trial. Allergy. 2005 Apr;60(4):494-500. doi: 10.1111/j.1398-9995.2004.00514.x. PMID 15727582
- [Background] Bonini S, Bonini S, Lambiase A, Marchi S, Pasqualetti P, Zuccaro O, Rama P, Magrini L, Juhas T, Bucci MG. Vernal keratoconjunctivitis revisited: a case series of 195 patients with long-term followup. Ophthalmology. 2000 Jun;107(6):1157-63. doi: 10.1016/s0161-6420(00)00092-0. PMID 10857837
- [Background] Leonardi A. Vernal keratoconjunctivitis: pathogenesis and treatment. Prog Retin Eye Res. 2002 May;21(3):319-39. doi: 10.1016/s1350-9462(02)00006-x. PMID 12052387